CLINICAL TRIAL: NCT00437489
Title: A 16 Week Open-Label Outpatient, Randomized, Parallel Study Assessing The Impact Of Two Different Initial Dose Prescriptions For Dry Powder Inhaled Insulin (Exubera®) On Glycemic Control In Patients With Type 2 Diabetes Mellitus Who Are Poorly Controlled On A Combination Of Two Or More Oral Agents.
Brief Title: A Clinical Trial Comparing The Efficacy And Safety Of 2 Different Initial Dose Prescriptions For Exubera.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This protocol was terminated not for safety reasons, but because Pfizer decided to return the worldwide rights for Exubera to Nektar, on 18 October 2007.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2171086
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Results first posted 2009-03-06 (Estimated); Last update posted 2009-05-11 (Estimated); Status verified 2009-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exubera

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Drug: Inhaled Human Insulin (Exubera)
- Experimental (Experimental)
  Interventions: Drug: Inhaled Human Insulin (Exubera)

INTERVENTIONS:
Drug: Inhaled Human Insulin (Exubera) — Initial dose (mg) as per weight based formula = 0.05 x body weight (kg) TID
  Arms: Control
Drug: Inhaled Human Insulin (Exubera) — Initial dose of 1mg TID of inhaled human insulin
  Arms: Experimental

SUMMARY:
The primary objective of this study is to assess whether a simple initial dose prescription of inhaled insulin (Exubera) achieves glycemic control (HbA1c) after 16 weeks that is non-inferior compared to the standard weight-based formula.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus Type 2
* Currently treated with at least 2 oral anti-diabetic agents

Exclusion Criteria:

* Severe Asthma, severe COPD
* Smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- Pfizer Investigational Site, Hong Kong, Hong Kong
- Pfizer Investigational Site, Karachi, Sindh, Pakistan
- Philippines (5):
  - Pfizer Investigational Site, Makati
  - Pfizer Investigational Site, Marikina City
  - Pfizer Investigational Site, Pasay
  - Pfizer Investigational Site, Pasig
  - Pfizer Investigational Site, Quezon City
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2171086&StudyName=A%20Clinical%20Trial%20Comparing%20The%20Efficacy%20And%20Safety%20Of%202%20Different%20Initial%20Dose%20Prescriptions%20For%20Exubera.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five centers in the Philippines, 2 centers in Singapore, 1 center in Hong Kong, and 1 center in Pakistan enrolled subjects.
Pre-assignment Details: As a result of Pfizer's decision (18Oct2007) to return the worldwide rights for Exubera (insulin human [rDNA origin]) Inhalation Powder) to Nektar, from which Pfizer licensed inhaled insulin technology, it was decided to terminate this study before it had recruited targeted number of subjects and followed them for the per protocol specified period.
Groups:
- Exubera Dose of 1mg Three Times Daily (TID): Subjects in Group A self-administered 1 mg Exubera TID before each meal (breakfast, lunch, and dinner)
- Exubera Dose (mg) as Per Weight Based Formula TID: Group B self-administered a dose of Exubera that was determined by the body weight-based formula = 0.05 x body weight (kg) TID.
Period: Overall Study
Arm/Group | Exubera Dose of 1mg Three Times Daily (TID) | Exubera Dose (mg) as Per Weight Based Formula TID
Started | 25 | 24
Completed | 2 (2 subjects completed prior to study termination.) | 2 (2 subjects completed prior to study termination.)
Not Completed | 23 | 22
Not completed — Study terminated by sponsor | 23 | 21
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exubera Dose of 1mg Three Times Daily (TID) | Exubera Dose (mg) as Per Weight Based Formula TID | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Customized [Number; unit: participants]
  <18 years | 0 | 0 | 0
  18 - 44 years | 3 | 5 | 8
  45 - 64 years | 20 | 17 | 37
  >= 65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 6 | 7 | 13

OUTCOME MEASURES:

1. Secondary Outcome: Fasting Plasma Glucose, and Overall Absolute, Pre-meal, and Post-meal Blood Glucose Change From Baseline to Week 16 (LOCF)
Description: Mean change of fasting plasma glucose, and overall absolute (based on the mean of 7-point home blood glucose monitoring (HGM) values), pre- and post-meal blood glucose (based on the mean of pre- or post-meal HGM values). Change from pre- to post-meal blood glucose based on the mean of difference of pre-meal HGM values from post-meal HGM values.
Time Frame: From baseline to week 16
Population: FAS - descriptive statistics were produced using LOCF for Week 16, therefore all subjects are included in the Week 16 data.
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Exubera Dose of 1mg Three Times Daily (TID) | Exubera Dose (mg) as Per Weight Based Formula TID
Number analyzed (Participants) | 25 | 24
mmol/l
  Fasting plasma glucose | -1.8 (2.36) | -2.9 (5.62)
  Overall absolute blood glucose | -2.5 (3.62) | -4.3 (4.20)
  Pre-meal blood glucose | -1.7 (3.58) | -3.3 (4.05)
  Post-meal blood glucose | -4.1 (3.78) | -5.5 (4.28)
  Change from pre-meal to post-meal blood glucose | -2.5 (2.14) | -2.1 (2.96)

2. Primary Outcome: Change in HbA1c From Baseline
Description: Mean change of hemoglobin A1c (HbA1c %) from baseline to week 16
Time Frame: From baseline to week 16
Population: Full analysis set (FAS) population - descriptive statistics were produced using last observation carried forward (LOCF) for Week 16, therefore all subjects are included in the Week 16 data.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Exubera Dose of 1mg Three Times Daily (TID) | Exubera Dose (mg) as Per Weight Based Formula TID
Number analyzed (Participants) | 25 | 24
Percent | -1.9 (1.56) | -2.0 (1.17)

3. Secondary Outcome: Number of Subjects Who Experienced Hypoglycemia and Nocturnal Hypoglycemia
Description: Cumulative Number Subjects Who Experienced Hypoglycemia & Nocturnal Hypoglycemia. Hypoglycemia:1)Clinical picture includes prompt resolution with food intake, subcutaneous glucagon, or intravenous glucose, 2)blood glucose check showing glucose <3.27 mmol/L (59 mg/dl), 3)glucose measurement of 2.7 mmol/L (49 mg/dl) or less, with or without symptoms.
Time Frame: week 16
Population: FAS Population - Descriptive statistics were produced using LOCF for Week 16, therefore all subjects are included in the Week 16 data.
Measure: Number; unit: participants
Arm/Group | Exubera Dose of 1mg Three Times Daily (TID) | Exubera Dose (mg) as Per Weight Based Formula TID
Number analyzed (Participants) | 25 | 24
participants
  Hypoglycemia | 12 | 5
  Nocturnal hypoglycemia | 2 | 2

4. Secondary Outcome: Hypoglycemia Event Rate Per Month
Description: Monthly event rate was calculated as the daily event rate multiplied by 30, and the daily event rate was calculated as the total number of events divided by the days in study up to the specified timepoint (ie, Week 4 or Week 16).
Time Frame: up to week 4 or 16
Population: FAS Population
Measure: Mean (Standard Deviation); unit: event rate per month
Arm/Group | Exubera Dose of 1mg Three Times Daily (TID) | Exubera Dose (mg) as Per Weight Based Formula TID
Number analyzed (Participants) | 25 | 24
event rate per month
  up to week 4 (GrpA:n=8, GrpB:n=4) | 3.3 (3.3) | 8.3 (9.1)
  up to week 16 (GrpA:n=12, GrpB:n=5) | 2.4 (2.4) | 2.5 (1.3)

ADVERSE EVENTS:
Arm/Group | Exubera Dose of 1mg Three Times Daily (TID) | Exubera Dose (mg) as Per Weight Based Formula TID
Serious Adverse Events (participants affected / at risk) | 2 | 0
Other Adverse Events (participants affected / at risk) | 17 | 15
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Exubera Dose of 1mg Three Times Daily (TID) | Exubera Dose (mg) as Per Weight Based Formula TID
Blood pressure inadequately controlled (Vascular disorders) | 1/25 | 0/24
Pelvic Instability at the Lumbar Spine (Musculoskeletal and connective tissue disorders) | 1/25 | 0/24
Diabetic Neuropathy (Nervous system disorders) | 1/25 | 0/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4.1% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Exubera Dose of 1mg Three Times Daily (TID) | Exubera Dose (mg) as Per Weight Based Formula TID
Eye disorders (Eye disorders) | 2/25 | 1/24
Gastrointestinal disorders (Gastrointestinal disorders) | 4/25 | 2/24
General disorders and administration site conditions (General disorders) | 5/25 | 6/24
Infections and infestations (Infections and infestations) | 3/25 | 1/24
Metabolism and nutrition discorders (Metabolism and nutrition disorders) | 12/25 | 5/24
Nervous system disorders (Nervous system disorders) | 10/25 | 6/24
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3/25 | 3/24
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 4/25 | 3/24
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0/25 | 2/24

LIMITATIONS AND CAVEATS:
As a result of Pfizer's decision (18Oct2007) to return the worldwide rights for Exubera (insulin human [rDNA origin]) Inhalation Powder) to Nektar, from which Pfizer licensed inhaled insulin technology, it was decided to terminate this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.